CLINICAL TRIAL: NCT00162760
Title: Treatment of Idiopathic Pulmonary Fibrosis With Thalidomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG00519
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2007-10

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The goal of this study is to determine whether thalidomide can stop the progression of fibrosis in IPF.

The primary objective of this study is to determine the safety, feasibility and efficacy of 400 mg of thalidomide administered daily for one year in patients with idiopathic pulmonary fibrosis (IPF) who have failed or are not candidates for treatment with corticosteroids and/or cytotoxic drugs.

The study population will consist of patients with biopsy-proven moderate to severe IPF who have failed or are not candidates for standard therapy with corticosteroids and/or cytotoxic drugs.

DETAILED DESCRIPTION:
This is an unmasked Phase II, safety and efficacy trial of subjects with biopsy-proven IPF who have failed or are not candidates for standard therapy with corticosteroids and/or cytotoxic drugs. The study doctors are interested in studying the effects of the oral drug Thalomid(R) on IPF. Thalomid(R) (thalidomide) is an approved medication for Hansen's disease (leprosy). It is know to have anti-inflammatory effects and effects on fibrosis. It is hoped that Thalomid(R) may prevent progression of IPF.

Thalidomide is investigational for this use, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) for the treatment of IPF.

The age range for this study is 50-80 years, inclusive. There are 6 visits over the 12 month period. These visits include physical exams, pregnancy tests (if applicable), several symptom scales and questionnaires about your pulmonary fibrosis, pulmonary function testing, x-rays,peripheral nerve testing, and blood tests including arterial blood gas measurements. You will be given the medication in capsule form every 28 days for a year. There is a set schedule for increasing the doses of the thalidomide every 2 weeks until it reaches the 400 mg. dose that is being studies. A stool softener is also provided for each participant.

All subjects must read, sign and follow a manual of precautions prepared by Celgene, the manufacturer of Thalomid(R), before enrolling in this study. This manual, containing the S.T.E.P.S.(R) precautions, will be given to all participants.

This study is being conducted at the Johns Hopkins Medical Institutions located in Baltimore, Maryland.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history consistent with IPF for greater than or equal to 3 months duration and less than 5 years.
* Documented IPF with UIP on histologic examination of surgical lung biopsy confirmed by study physician (RT).
* High resolution CT (HRCT) of chest consistent with IPF (bibasilar reticular abnormalities with minimal ground glass opacities) as determined by study physician (KMH).
* Failure to have >/= 10% increase in FVC on prior adequate treatment with corticosteroids and/or cytotoxic drugs, or intolerance to these drugs precluding use.
* FVC >/= 40% and </= 90% predicted at screening.
* DLCo >/= 25% predicted at screening
* Oxygen saturation >/= 88% on room air or </= 2L oxygen at screening.
* Age 50-80 inclusive
* Ability to understand and sign informed written consent form and comply with study guidelines

Exclusion Criteria:

* Known etiology of ILD (e.g. sarcoid, hypersensitivity pneumonitis, BOOP etc.)
* Clinically significant toxic or environmental exposure to respiratory irritants (e.g. drugs, asbestosis, radiation etc.)
* Diagnosis of collagen vascular disease.
* Obstruction on PFTs, defined as FEV1/FVC < 0.6.
* Active infection
* End stage coronary artery disease, congestive heart failure or cor pulmonale
* History of significant peripheral vascular disease
* History of peripheral neuropathy
* History of clinically significant obstructive sleep apnea
* History of poorly controlled diabetes
* Pregnant or lactating women
* Abnormal laboratories as defined as: WBC < 2300/mm3, HCT < 30% or >55%, PLT < 100k/mm3. creatinine >1.5, AST or ALT > 3x normal, total bilirubin > 1.5.
* Current enrollment in another protocol for IPF
* Prednisone use >15 mg a day in 4 weeks prior to starting trial.
* Cytotoxic drugs (cyclophosphamide, azathioprine, colchicines, cyclosporine, interferon-gamma) 6 weeks prior to screening.
* Patients requiring chronic narcotic analgesic.
* Patients unable to give informed consent.
* Patients unable to comply with the requirements for the trial.
* Patients with known allergy/intolerance to thalidomide;
* Patients with a predicted life expectance less than 6 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2003-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety, feasibility and efficacy of 400 mg of thalidomide administered daily for one year in patients with IPF who have failed or are not candidates for treatment with corticosteroids and/or cytotoxic drug.

SECONDARY OUTCOMES:
The efficacy of thalidomide in preventing progressive pulmonary fibrosis and clinical deterioration measured objectively with changes in PFTs and radiographs as well as with dyspnea scales and quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen R Horton, M.D., Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: Johns Hopkins Pulmonary & Critical Care Medicine website — http://www.hopkinsmedicine.org/pulmonary/
- See also: Pulmonary Fibrosis Foundation — http://www.pulmonaryfibrosis.org/